CLINICAL TRIAL: NCT03144752
Title: Optimizing Clinical Screening and Management of Maternal Mental Health: Predicting Women at Risk for Perinatal Depression
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108271; NAPND0001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Participants between 8 to 14 weeks gestation: Cohort 1 will include female participants who present for the first prenatal visit which takes place between Weeks 8 and 14 at maternity practices associated with University of North Carolina (UNC) Women's Care. Biomarkers, medical and psychiatric history, and psychosocial measures will be evaluated and utilized in developing a predictive risk algorithm for perinatal depression.
- Cohort 2: Participants between 15 to 36 weeks gestation: Cohort 2 will include female participants enrolled at various points in their pregnancy from Week 15 up through 36 weeks gestation. Biomarkers, medical and psychiatric history, and psychosocial measures will be evaluated and utilized in developing a predictive risk algorithm for perinatal depression.

SUMMARY:
The purpose of this study is to determine if medical, biological, psychological, and social risk factors can be used to develop algorithms that will predict perinatal depression (PND). Data capture will include baseline participant medical, psychological and family history, blood biomarkers, and psychosocial assessments.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be English-speaking and able to understand and follow clinician/researcher/provider recommendations
* Participants must be able to read and comprehend written communications (English) and physically able to complete electronic patient-reported outcome (ePRO) assessments
* Participants must have access to a personal smartphone or a computer and an active personal email address for which they are willing to use for data collection
* Each participant must sign an informed consent form (ICF) indicating that she understands the purpose of and procedures required for this study and is willing to participate in and comply with all procedures in the study
* Participant must be willing and able to have blood draws and to complete the self-reported assessments via mobile electronic device during the study

Exclusion Criteria:

* Participant is not English speaking
* Lifetime mood disorder other than major depressive disorder (MDD) (example [e.g.], bipolar I) or anxiety disorder
* Lifetime psychotic disorder (eg, schizophrenia, schizoaffective disorder)
* Lifetime alcohol or illicit substance dependence (moderate-severe)
* Current Post-traumatic Stress Disorder (PTSD), significant alcohol or illicit drug use (Ethanol [ETOH]/nonprescription drug use) within 12 months greater than or equal to (>=)occasional use

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Approximately 300 pregnant women seeking maternal healthcare services in a department of Obstetrics and Gynecology at the University of North Carolina health center will be observed for perinatal depression.
Sampling Method: Non-Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2019-05-05 (Actual)

PRIMARY OUTCOMES:
Biomarker Assessment for Perinatal Depression | Up to Visit 3 (Weeks 36-40 of gestation)
  Blood samples will be collected to evaluate biomarkers for perinatal depression.
Medical and Psychiatric History | Visit 1 (anywhere between Weeks 8-36 of gestation)
  Participants will be asked to complete medical and psychiatric history questionnaire during their 1st visit.
Maternity Social Support Scale (MSSS) Score | Up to 24-26 weeks postpartum
  This is a brief 6 item questionnaire used a 5 level Likert type scale to assess perceived social support during the prenatal period. The score on each item within this scale (ranging from 1 to 5) is summarized according to the origin of support (eg, support from family/friends and support from partner). The total score is 30 with classified social support in to three categories; high social support (for scores 24-30), medium social support (18-23) and low social support (below 18) categories. High total score indicates increased perceived support.
Edinburgh Postnatal Depression Scale (EPDS) | Up to 24-26 weeks postpartum
  The EPDS is a self-administered scale that indicates how the mother has felt during the previous week. The scale consists of 10 questions. Responses are scored 0, 1, 2, or 3 according to increased severity of the symptom. The total score is determined by adding together the scores for each of the 10 items. The EPDS total score ranges from 0 to 30. A score of greater than (>)9 is indicative of perinatal major depression.
Perceived Stress Scale (PSS) | Up to 24-26 weeks postpartum
  The Perceived Stress Scale (PSS) measures the degree to which situations in one's life are appraised as stressful. The questionnaire asks the client about their perceived stress and their feelings and thoughts during the last month. The scale has ten questions asking respondents to circle a number between 0 and 4: 0 = Never, 1 = Almost Never, 2 = Sometimes, 3 = Fairly Often and 4 = Very Often. The range of possible score is from 0 to 40. Scores around 13 are considered average. Scores of 20 or higher are considered to be indicative of high stress levels.
State-trait Anxiety Inventory (STAI) | Up to 24-26 weeks postpartum
  The State-Trait Anxiety Inventory (STAI) is a measure of trait and state anxiety. STAI contains 20 items for assessing trait anxiety and 20 items for state anxiety. State anxiety items include: "I am tense; I am worried" and "I feel calm; I feel secure." Trait anxiety items include: "I worry too much over something that really doesn't matter" and "I am content; I am a steady person." All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Scores may range from 20 to 80 with higher scores indicating greater state anxiety.
Obsessive Compulsive Inventory - Revised (OCI-R) | Up to 24-26 weeks postpartum
  The OCI-R, a shortened version of the Obsessive-Compulsive Inventory, assesses symptoms of Obsessive Compulsive Disorder (OCD). The measure consists of 18 items (e.g. "I frequently have get nasty thoughts and have difficulty in getting rid of them"). On a five point scale, respondents rate how distressed or bothered they have been in the past month by the symptom described, with responses ranging from "Not at all" to "Extremely." Scores are generated by adding the item scores. Total possible score range 0 to 72, scores at or above 21 indicating the likely presence of OCD.
Patient-Reported Outcomes Measurement Information System (PROMIS)- Pain Interference | Up to 8-9 weeks postpartum
  Self-reported changes in the levels of pain as measured by the PROMIS Pain Interference Scale. PROMIS-PI scores provided substantial information across levels of pain. The scale for adults in the general population is available in both a 41 item long-form computer adaptive version and a 4 item short form which will be used in this study. Each item is based on experiences in the last seven days before administering the questionnaire. It uses a 5-point rating scale (1-"not at all" to 5-"very much"), with higher scores indicating more pain interference.
PROMIS-Sleep Disturbance | Up to 24-26 weeks postpartum
  The PROMIS-Sleep Disturbance (PROMIS-SD) is used to asses self-reported perceptions of sleep quality, sleep depth and restoration associated with sleep. The full PROMIS- SD includes 27 with each item is based on a 7-day recall period and assessed on a 5 level Likert-type scale. The 8 item short form will be used in this study, in which responses are scored 1 to 5 for each item. A higher score on 5 of the 8 items reflects a worse outcome, whereas a higher score on 3 items reflects an improved outcome; therefore, the directionality of the 8 item scores are first synchronized prior to calculation of the total raw score. To find the total raw score for a short form with all questions answered, sum the values of the response to each question. For example, for the adult 8-item form, the lowest possible raw score is 8; the highest possible raw score is 40. PROMIS scores are presented as T-scores. Higher T-scores represent more of the concept being measured (sleep disturbance).
PROMIS-Sleep Related Impairment | Up to 24-26 weeks postpartum
  The Patient Reported Outcomes Measurement Information System (PROMIS)Sleep Related Impairment bank is a 16 item computer adaptive test bank that focuses on perceptions of alertness, sleepiness, and tiredness during usual waking hours. Each item is based on a seven day recall period and assessed on a 5 score for a short form with all questions answered, sum the values of the response to each question. For example, for the adult 8-item form, the lowest possible raw score is 8; the highest possible raw score is 40. To find the total raw score for a short form with all questions answered, sum the values of the response to each question. For example, for the 8-item form, the lowest possible raw score is 8; the highest possible raw score is 40. PROMIS scores are presented as T-scores. Higher T-scores represent more of the concept being measured (sleep related impairment).
PROMIS-Self Efficacy | Up to 24-26 weeks postpartum
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Self-Efficacy for Managing Emotions is designed for adults with at least 1 chronic health condition. The items are not focused on one specific condition but are designed to universally measure one's current level of confidence to manage emotional symptoms such as anxiety, depression, helplessness, discouragement, frustration, disappointment and anger. The instrument has a 25 item computer adaptive test form and 2 short forms: an 8 item and a 4 item. Each question has 5 response options ranging in value from 1 to 5. To find the total raw score for a short form with all questions answered, sum the values of the response to each question. For example, for the 8-item form, the lowest possible raw score is 8; the highest possible raw score is 40. PROMIS scores are presented as T-scores. Higher T-scores represent more of the concept being measured (self efficacy).
Patient Health Questionnaire-2 (PHQ-2) | Up to 24-26 weeks postpartum
  The Patient Health Questionnaire-2 (PHQ-2) is a 2-item Brief Depression Screening Instrument. It inquires about the frequency of depressed mood and anhedonia over the past 2 weeks, scoring each as 0 ("not at all") to 3 ("nearly every day"). It ranges from 0-6, where higher score means higher depressive symptoms.
Perinatal Post-traumatic Stress Disorder (PTSD) Questionnaire - Modified (PPQ) | At 12-14 weeks postpartum
  The Perinatal Post-Traumatic Stress Disorder (PTSD) Questionnaire (PPQ) is a 14-item measure assessing post-traumatic symptoms related to the childbirth experience, including intrusiveness or re-experiencing, avoidance behaviors and hyperarousal or numbing of responsiveness. The PPQ also contains one item pertaining to feelings of guilt. Response options were modiﬁed from the original dichotomous scale to a ﬁve-level likert scale (scored 0 to 4). Mothers were instructed to provide responses that reﬂected their experience during the targeted time frame (4 to18 months postpartum). The total possible score on the modiﬁed PPQ ranged from 0 to 56. A score of 19 or higher on the PPQ indicates clinically significant distress that merits referral of the mother to a mental health care professional.
Generalized Anxiety Disorder-7 (GAD-7) | Up to 24-26 weeks postpartum
  The GAD-7 is a self-reported questionnaire for screening and measurement of severity of generalized anxiety disorder (GAD). This questionnaire has 7 items which measure the severity of various signs of GAD over the past 2 weeks according to the reported response categories with assigned points - "not at all" (0 points), "several days" (1 point), "more than half the days" (2 points), and "nearly every day" (3 points). Total score=sum of all 7 items; ranges from 0 to 21; Higher score=greater level of anxiety).
Pregnancy-Unique Quantification of Emesis and Nausea - Modified (PUQE) | Up to 24-25 weeks
  The modified version of the Pregnancy-Unique Quantification of Emesis and Nausea (modified-PUQE) provides global nausea and vomiting of Pregnancy (NVP) severity index. The modified-PUQE is a three-item questionnaire with each item having a 5 level Likert type scale (1 to 5, increasing in severity). The total score is the sum of replies to the 3 items and rated from 3 (no symptoms) to 15 (most severe). A score of 7 to 12 indicates moderate NVP and a score greater than 13 indicates severe NVP.
Infant Feeding Intentions Scale (IFI) | At 24-25 weeks
  The Infant Feeding Intentions (IFI) scale was developed to meet the need in breastfeeding behavior studies for quantitative measure of maternal breastfeeding intentions. This is a 5 item scale that probes strength of intentions to initiate breastfeeding. Total score ranges from 0 to 16. Higher score means higher intention to breastfeed exclusively.
Neonatal Breastfeeding Questionnaire | At 5-9 days postpartum
  The questions used to assess breastfeeding behavior immediately post-delivery are adapted from Infant Feeding Practices Study II (IFPS II). The Neonatal Questionnaire was sent to the mother when her infant is approximately 3 weeks old. This questionnaire examined factors that commonly occur near the time of the birth and that affect infant feeding choices. This study will use 3 of their face valid questions to assess if the new mother has tried to breastfeed, if so, how long it took for her milk to produce, and if she is still breastfeeding.
Postnatal Breastfeeding Questionnaire | At 24-26 weeks postpartum
  The questions used to assess longitudinal breastfeeding behavior post-delivery are also adapted from Infant Feeding Practices Study II (IFPS II). The Postnatal Questionnaires consist of various combinations of 8 modules that were mailed to the mother approximately monthly from the time her infant is 2 months through 12 months of age. A 4 question subset of the breastfeeding questionnaire will be used in this study to evaluate continued breastfeeding practices and reasons to begin using formula or to stop breastfeeding.

SECONDARY OUTCOMES:
Incidence of Perinatal Depression (PND) | Up to 60 weeks
  Incidence of PND will be assessed at different time points, including those participants who are already depressed at baseline and both antenatal and postpartum depression onset in a real world population of pregnant women seeking health care.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States